CLINICAL TRIAL: NCT04392765
Title: The Efficacy of Intra-oral Neuromuscular Stimulation Training on Snoring in Individuals With Primary Snoring or Mild Sleep Apnoea - A Multi Centre Trial
Brief Title: Efficacy of Intra-oral Neuromuscular Stimulation Training on Snoring and Mild Sleep Apnoea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Signifier Medical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: eXciteOSA Multicentre
Record Dates: First submitted 2020-05-11; First posted 2020-05-19 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Snoring; Sleep Apnea, Obstructive
MeSH Terms: conditions — Snoring; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Therapy arm (Other): Six week use of eXciteOSA device. Once daily for 20 minutes.
  Interventions: Device: eXciteOSA

INTERVENTIONS:
Device: eXciteOSA — eXciteOSA transoral neurostimulation device

SUMMARY:
It has been shown that a common cause for snoring and throat obstruction (obstructive sleep apnoea (OSA)) is excessive loss of muscle tone in the throat when the investigators go to sleep. This results in the partial collapse of the throat (snoring) or complete collapse (OSA) during sleep.

45% of the male population snore. Sleep apnoea affects 4 to 6% of the population and is associated with increased incidence of raised blood pressure, heart attacks and strokes. Although there are several lifestyle practices associated with snoring such as smoking, obesity and drinking, a significant proportion of people may snore despite not being associated with these.

A solution to this issue is to improve the muscle tone of the throat so that it doesn't collapse so easily. Several studies have shown that certain types of throat exercises can help reduce snoring. Further studies have also shown that using electrical stimulation to exercise the tongue muscles has the same effect.

From this, doctors in the United Kingdom (UK) have developed a new type of device, eXciteOSA, that allows a more accurate and comfortable way of delivering this energy to exercise the tongue muscles. The device works by stimulating the tongue muscles during the day so that the tongue is less likely to collapse during sleep. It is a form of "workout" for the tongue and like other physical exercise regimes, it needs to be repeated regularly for a few weeks to take effect.

The aim of this study is to see if the eXciteOSA device is as effective as the previous methods and if it can reduce snoring and improve sleep quality.

This will be achieved by participants using the eXciteOSA once daily for a six week period. A two night sleep study with watchPAT along with a polysomnography will be completed before and after the therapy to compare results. Questionnaires on sleep quality and quality of life will also be completed pre and post therapy.

DETAILED DESCRIPTION:
Study Design: Phase IV prospective, multi-centre post-market surveillance study.

Each site will follow the pre-determined study protocol, collecting endpoint relevant data which will then be analysed according to the methods outlined in this statistical analysis plan (SAP).

In brief, participants will proceed through three phases of the trial. The pre-trial phase collects data on the pre therapy state of the participant, after which they will enter the therapy phase where they use the device once daily for the required period whilst continuing to record the required data. The participant will stop using the device at the end of this stage and have a follow up phase during which trial indices will continue to be recorded.

The eXciteOSA transoral neurostimulation device is a home use device controlled by a mobile app. Its primary indication is for use in snoring in primary snorers or individuals with mild sleep apnoea.

It is reusable device that produces muscular stimulation via electrodes integrated into a mouthpiece used by the candidate. The product will be supplied be Signifier Medical Technologies ltd. The eXciteOSA device comes in a black box which contains the control unit, mouthpiece, universal serial bus (USB) cable and the instructions for use. Only the supplied products should be used together. Use of the product should be discontinued if it appears damaged in any way. The mouthpiece is connected to the control unit via a USB port and Bluetooth connection is established between the control unit and the app.

The device is to be used whilst awake, once daily for 20 minutes. The app automatically times the session and terminates it once completed. The therapy consists of a series of pulse bursts with the basic characteristic of 6 secs burst and 4 seconds rest. During the 20 mins therapy period the pulse frequency will change every 5 mins in a defined sequence. The intensity of the pulses can be controlled be the participant using the app, from a scale of 1 to 15. Patients should select the highest level they can tolerate without any discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial
* Male or female, aged 18 years or above
* AHI 5-15/hr as confirmed by polysomnography performed for screening purposes
* Snoring complaints for >6 months
* In possession of a smartphone (to use the application)

Exclusion Criteria:

* BMI >35 kg/m2
* AHI >15/h, i.e. evidence of moderate to severe obstructive sleep apnoea (OSA) from polysomnography
* Symptomatic nasal pathology i.e. septal deviation, nasal polyposis or chronic rhinosinusitis
* Tonsil Hypertrophy (Tonsil size - Grade 3 or greater)
* Tongue or lip piercing
* Pacemaker or implanted medical electrical devices
* Previous oral surgery for snoring
* Relevant facial skeletal abnormalities (i.e. syndromic facial deficiencies, severe micrognathia etc.)
* Pregnancy or planned pregnancy
* Any criteria that, in the opinion of the investigator, would make the participant unsuitable for the study due to inability to complete required study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in sleep disordered breathing indices - Apnea Hypopnea Index (AHI) | Change between pre-therapy (day 0) and post therapy (day 49)
  To assess the efficacy of daytime trans-oral neuromuscular stimulation training on respiratory indices of Sleep disordered breathing (AHI)
Change in sleep disordered breathing indices - Oxygen Desaturation Index (ODI) | Change between pre-therapy (day 0) and post therapy (day 49)
  To assess the efficacy of daytime trans-oral neuromuscular stimulation training on respiratory indices of Sleep disordered breathing (ODI)
Change in Objective snoring pre and post therapy | Change between pre-therapy (day 0) and post therapy (day 49)
  To assess the efficacy of daytime trans-oral neuromuscular stimulation training on objective snoring in Sleep disordered breathing (% snoring at 40, 45 and 50dB)

SECONDARY OUTCOMES:
Comparison of sleep quality questionnaires at start and end of therapy - Pittsburgh Sleep Quality Index (PSQI) | Change between pre-therapy (day 7) and post therapy (day 49)
  To assess the efficacy of daytime trans-oral neuromuscular stimulation training on snoring sleep quality.
Comparison of sleep quality questionnaires at start and end of therapy - Epsworth Sleepiness Score (ESS) | Change between pre-therapy (day 7) and post therapy (day 49)
  To assess the efficacy of daytime trans-oral neuromuscular stimulation training on snoring sleep quality.
Comparison of visual analogue scale (VAS) of snoring reported by partner | Change between pre-therapy (day 7) and post therapy (day 49)
  To assess the efficacy of daytime trans-oral neuromuscular stimulation training on snoring reported by sleep partner
Comparison of quality of life questionnaires at start and end of therapy - EQ-5D-5L | Change between pre-therapy (day 7) and post therapy (day 49)
  To assess the efficacy of daytime trans-oral neuromuscular stimulation training on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Zayni, Study Director — Signifier Medical Technologies
Locations (6):
- Canada (2):
  - Vancouver Hospital, Vancouver, British Columbia
  - McGill University Health Centre, Montreal
- Advanced Sleep Research GMBH, Berlin, Germany
- OLVG, Amsterdam, Amsterdam, Netherlands
- Spain (2):
  - Clínica Universidad de Navarra, Pamplona, Pamplona
  - Hospital Universitario Doctor Peset, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No